CLINICAL TRIAL: NCT02361203
Title: Exercise and Virtual Reality Exposure Therapy for Acrophobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jolene Jacquart, Graduate Student, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2014-12-0037
Record Dates: First submitted 2015-01-29; First posted 2015-02-11 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Fear of Heights
MeSH Terms: conditions — Acrophobia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Exercise (No Intervention)
- Exercise Pre (Experimental): 30 minutes of aerobic exercise before exposure therapy
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 30 minutes of aerobic exercise on a treadmill at 80% of participant's heart rate reserve.
  Arms: Exercise Pre

SUMMARY:
The purpose of this study is to determine whether aerobic exercise can enhance the effects of exposure therapy treatment for fear of heights.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 25
* Speaks English fluently
* Score of 80 or higher on the Acrophobia Questionnaire
* SUDS rating of 50 or higher on the Behavioral Avoidance Test or complete refusal to comply with instructions due to intensity of fear
* Passes the Physical Activity Readiness Questionnaire-Plus

Exclusion Criteria:

* Hearing or visually impaired
* Currently receiving exposure-based treatment for acrophobia
* Able to remain on floor 20 for 30 seconds during BAT with a SUDS rating < 50

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Fear scores | 7 (+/- 3) days after exposure therapy
  Change in fear scores using subjective units of distress will be assessed.
Perceived threat likelihood scores | 7 (+/- 3) days after exposure therapy
  Change in the perception of threat likelihood on a scale from 1-5 will be assessed.

SECONDARY OUTCOMES:
Skin conductance fluctuations | 7 (+/- 3) days after exposure therapy
  Changes in skin conductance fluctuations will be assessed.
Heart rate fluctuations | 7 (+/- 3) days after exposure therapy
  Heart rate fluctuations will be assessed.
Acrophobia Severity | 14 (+/- 3) days after exposure therapy
  Change in score on the Acrophobia Questionnaire
Attitudes Toward Heights | 14 (+/- 3) days after exposure therapy
  Change in score on the Attitudes Toward Heights Inventory
Clinical Global Improvement | 14 (+/- 3) days after exposure therapy
  Change in score on the Clinical Global Improvement Scale

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Smits, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States